CLINICAL TRIAL: NCT05999344
Title: Exploring Intoxication During Acute Alcohol and Cannabis Concentrate Co-Administration: A Focus on Cannabinoid Content and Order Effects
Brief Title: Alcohol and Cannabis Concentrates Co-Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Institute of Cannabis Research, Colorado State University Pueblo (Unknown); Colorado State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2161
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Alcohol Use Disorder; Cannabis Use
Keywords: alcohol; cannabis; polysubstance use; psychomotor impairment; cannabis concentrates
MeSH Terms: conditions — Alcoholism; Marijuana Abuse; Psychomotor Disorders | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol before Cannabis (Experimental): Participants are randomly assigned to receive the standardized alcohol dose during the experimental session prior to going inside their residence to self-administer their preferred cannabis concentrate product.
  Interventions: Other: commercially available alcohol administered prior to commercially available cannabis
- Cannabis before alcohol (Experimental): Participants are randomly assigned to go inside their residence to self-administer their preferred cannabis concentrate product and then receive the standardized alcohol dose.
  Interventions: Other: commercially available cannabis administered prior to commercially available alcohol

INTERVENTIONS:
Other: commercially available cannabis administered prior to commercially available alcohol — Self administration of cannabis prior to researcher administered alcohol
  Arms: Cannabis before alcohol
Other: commercially available alcohol administered prior to commercially available cannabis — Researcher administered alcohol prior to self-administration of cannabis
  Arms: Alcohol before Cannabis

SUMMARY:
The goal of this study is to learn about the effects of combining alcohol with cannabis concentrate products which contain high levels of THC. The main question[s] it aims to answer are, 1) How does the order in which someone consumes THC and alcohol in a given co-use session impact outcomes such as blood alcohol level, heart rate or subjective drug effects, and 2) how does THC percentage in cannabis influence outcomes following alcohol and cannabis co-administration. Participants will be scheduled for our mobile lab to come to their residence. During the session, they will:

* consume a standardized dose of alcohol as well as use their own preferred cannabis concentrate product.
* they will then remain in our mobile lab for about 4 hours and complete some surveys as well as do some cognitive tasks on an iPad every 30 minutes.
* They will also have their blood drawn three times throughout the session, and will periodically be asked to blood into a breathalyzer to measure blood alcohol level.

Researchers will compare people who use alcohol prior to cannabis to those who use cannabis prior to alcohol to determine whether order of use impacts outcomes.

DETAILED DESCRIPTION:
Individuals who drink alcohol commonly report co-using cannabis, and the increasing availability of new formulations of highly potent cannabis products on the legal market means that alcohol is likely being combined with cannabis products that contain high levels of delta-9-tetrahydrocannabinol (THC). There is limited existing research on the acute effects of cannabis products containing high amounts of THC, such as cannabis concentrates, which often contain up to 90% THC. Existing laboratory data suggests that consuming alcohol and cannabis together (compared to alcohol alone) is associated with reduced BAC, delayed time to peak blood alcohol concentration (BAC), longer duration of intoxication, and increased subjective intoxication, but it is unknown how cannabis concentrates may interact with alcohol to influence these outcomes. There is also a lack of research regarding whether timing or order of use matters, though recent survey data from our group and others suggests that using alcohol before cannabis may confer additional risk compared to using cannabis prior to alcohol. The present study leverages a federally-compliant mobile laboratory design to explore the acute effects of self-administered cannabis concentrates alongside a standardized dose of alcohol. The investigators will recruit a community sample of individuals who regularly use alcohol and cannabis to participate study sessions in our mobile laboratory. The sessions will involve individuals consuming cannabis concentrates of their choice (that they acquire themselves) along with a standardized dose of alcohol. Half of the participants will use the alcohol before cannabis, and the other half will use the cannabis before alcohol. The investigators will measure intoxication and biological outcomes every 30 minutes for 4 hours. The investigators will also measure differences between those who used alcohol before cannabis and those who used cannabis before alcohol.

ELIGIBILITY:
Inclusion Criteria:

1. 21-65 years old,
2. Heavy drinkers (for men, >4 drinks in one occasion, or >14 drinks per week; for women, >3 drinks in one occasion, or >7 drinks per week)
3. Regular users of legal-market cannabis (at least 3x/week in past 3 months)
4. Have experience using cannabis concentrates within the last year
5. Willing to obtain a concentrate product of their choice for use in the study.

Exclusion Criteria:

1. Diagnosed with or seeking treatment for alcohol use disorder (AUD) or other substance use disorder (SUD)
2. Pregnant, breastfeeding or trying to become pregnant
3. Meet criteria for psychotic, bipolar or major depressive disorder with suicidal ideation, or history of these disorders
4. Current use of psychotropic (except anti-depressants) or steroid medications
5. Report illicit drug use in past 60-days or fail drug screen (drug screen tests for the presence of amphetamines, benzodiazepines, cocaine, THC, methamphetamine and opioids; only THC is allowed to be present in urine in order to be eligible to participate in the study
6. Major medical condition contraindicating alcohol and/or cannabis consumption (e.g., liver disease, heart disease, or being told by a doctor that it is unsafe to consume alcohol or cannabis due to a medical condition)
7. Have participated in another research study in the past 8 weeks.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Breath Alcohol Level (BrAC) | Baseline (pre ingestion) and every 30 minutes (post ingestion) for a total of 270 minutes (9 measures)
  Breath alcohol level will be measured using a breathalyzer repeatedly during the experimental session
Alcohol Urge Questionnaire (AUQ) | Baseline (pre ingestion) and every 30 minutes (post ingestion) for a total of 270 minutes (9 measures)
  The AUQ is a self-report measure of urge for alcohol and has been validated for real-time assessment of alcohol craving in the laboratory. The total score on the measure ranges from 0-48 where higher is worse
Heart Rate (HR) | Baseline (pre ingestion) and every 30 minutes (post ingestion) for a total of 270 minutes (9 measures)
  Heart rate (beats per minute) is measured using a finger pulse oximeter
ARCI Marijuana Scale | Baseline (pre ingestion) and every 30 minutes (post ingestion) for a total of 270 minutes (9 measures)
  The ARCI scale measures subjective responses to cannabis. total score ranges from 0-12 where higher is worse
DRUID Psychomotor Battery | Baseline (pre ingestion) and every 30 minutes (post ingestion) for a total of 270 minutes (9 measures)
  The DRUID is a mobile app that tests for cognitive and motor impairment, and has been shown to detect impairment related to alcohol and cannabis use. total score ranges from 0-100 where higher is worse.

SECONDARY OUTCOMES:
Blood-THC | Blood is drawn immediately prior to alcohol and cannabis consumption, again 60 minutes post alcohol administration start time, and again 240 minutes post alcohol start time
  We will quantify levels of THC in the blood before and after the participant uses their cannabis product
Biphasic Effects of Alcohol Scale (BAES) | Baseline (pre ingestion) and every 30 minutes (post ingestion) for a total of 270 minutes (9 measures)
  The BAES measures the stimulating and sedating effects of alcohol and is validated for use in laboratory settings. This scale produces a stimulation subscale (total score ranges from 0-70 where higher is more stimulated) and a sedation subscale (total score ranging from 0-70 where higher is more sedated)
Profile of Mood States (POMS) | Baseline (pre ingestion) and every 30 minutes (post ingestion) for a total of 270 minutes (9 measures)
  The POMS is a self-report rating scale that assesses state-level, distinct mood states. The POMS produces multiple subscales (Tension, depression, anger, fatigue, confusion, vigour, as well as a total mood disturbance scale)

CONTACTS AND LOCATIONS:
Overall Officials: Hollis C Karoly, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No